CLINICAL TRIAL: NCT03706547
Title: Clinical Study of Anti-CD19/BCMA Bispecific Chimeric Antigen Receptors (CARs) T Cell Therapy for Relapsed and Refractory Multiple Myeloma
Brief Title: Anti-CD19/BCMA Bispecific CAR-T Cell Therapy for R/R MM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peng Liu (Other)
Collaborators: Hrain Biotechnology (Unknown); Shanghai East Hospital (Other)
Responsible Party: Sponsor-Investigator, Peng Liu, Professor, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHZS-MM002
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma Progression
MeSH Terms: interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19/BCMA CAR-T cells (Experimental): 1. Chemotherapy with a classic combination with fludarabine and cyclophosphamide;
  2. Administration with anti-CD19/BCMA CAR-T cells in the BCMA-positive multiple myeloma patients.
  Interventions: Biological: anti-CD19/BCMA CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: anti-CD19/BCMA CAR-T cells — Retroviral vector-transduced autologous T cells to express anti-CD19 and anti-BCMA CARs
Drug: Fludarabine — 30mg/m2/d
Drug: Cyclophosphamide — 300mg/m2/d

SUMMARY:
The goal of this clinical trial is to study the feasibility and efficacy of anti-CD19/BCMA bispecific chimeric antigen receptors (CARs) T cell therapy for relapsed and refractory multiple myeloma.

DETAILED DESCRIPTION:
Primary Objectives

1. To determine the feasibility ad safety of anti-CD19/BCMA CAR-T cells in treating patients with BCMA-positive multiple myeloma.

Secondary Objectives

1. To access the efficacy of anti-CD19/BCMA CAR-T cells in patients with multiple myeloma.
2. To determine in vivo dynamics and persistency of anti-CD19/BCMA CAR-T cells.

ELIGIBILITY:
Inclusion Criteria:

* Expected survival > 12 weeks
* Diagnosis of Multiple Myeloma by IMWG updated criteria (2014)
* Pathology demonstrated that BCMA-poitive malignant plasma cells exited in bone marrow or plamacytoma
* Exited measurable lesions and in accordance with one of the following test indicators: serum M protein≥1 g/dl; urine M protein≥200 mg/24h; serum free light chain≥10 mg/dl; diagnosis of plasmacytoma by biopsy
* The criteria for relapsed and refractory multiple myeloma: patients previously received at least 3 different prior treatment regimens for multiple myeloma, including protein inhibitors (eg: Bortezomib), and immunomodulator (eg: Revlimid), and have disease progression in the past 60 days
* At least 90 days after stem cell transplantation
* Clinical performance status of ECOG score 0-2
* Creatinine≤2.0 mg/dl
* Bilirubin≤2.0 mg/dl
* The ALT/AST value is lower than 2.5-fold of normal value
* Accessible to intravenous injection, and no white blood cell collection contraindications
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 30 days after the CTL infusion. Male partner should use a condom
* 5mg/day dose of Prednisone or other equivalent steroid hormone drugs (eg: Dexamethasone) were not used for two weeks before apheresis and CAR-T infusion
* Able to understand and sign the Informed Consent Document.

Exclusion Criteria:

* Patients with symptoms of central nervous system
* Patients with second malignancies in addition to multiple myeloma
* Active hepatitis B or C, HIV infections
* Any other active diseases could affect the enrollment of this trial
* Long term use of immunosuppressive agents after organ transplantation, except currently receiving or recently received glucocorticoid treatment
* Patients with organ failure
* Women of child-bearing potential who are pregnant or breastfeeding during therapy, or have a planned pregnancy with 2 months after therapy
* A history of mental illness and poorly controlled
* Women of child-bearing potential who are not willing to practice birth control from the time of enrollment on this study and for 2 months after receiving the preparative regimen. Women of child bearing potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion
* Patients who are accounted by researchers to be not appropriate for this test
* Subjects suffering disease affects the understanding of informed consent or complying with study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-30 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 4.0 | 6 months
  Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 4.0

SECONDARY OUTCOMES:
Overall remission rate defined by the standard response criteria for myeloma for each arm | 8 weeks
  Overall remission rate defined by the standard response criteria for myeloma for each arm
Duration of CAR-positive T cells in circulation | 6 months
  Duration of CAR-positive T cells in circulation

CONTACTS AND LOCATIONS:
Overall Officials: Peng Liu, M.D. & Ph.D., Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Department of Hematology ,Fudan University Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] Child JA, Morgan GJ, Davies FE, Owen RG, Bell SE, Hawkins K, Brown J, Drayson MT, Selby PJ; Medical Research Council Adult Leukaemia Working Party. High-dose chemotherapy with hematopoietic stem-cell rescue for multiple myeloma. N Engl J Med. 2003 May 8;348(19):1875-83. doi: 10.1056/NEJMoa022340. PMID 12736280
- [Background] Hari PN, McCarthy PL. Multiple myeloma: future directions in autologous transplantation and novel agents. Biol Blood Marrow Transplant. 2013 Jan;19(1 Suppl):S20-5. doi: 10.1016/j.bbmt.2012.11.002. No abstract available. PMID 23290439
- [Background] Bruno B, Rotta M, Patriarca F, Mordini N, Allione B, Carnevale-Schianca F, Giaccone L, Sorasio R, Omede P, Baldi I, Bringhen S, Massaia M, Aglietta M, Levis A, Gallamini A, Fanin R, Palumbo A, Storb R, Ciccone G, Boccadoro M. A comparison of allografting with autografting for newly diagnosed myeloma. N Engl J Med. 2007 Mar 15;356(11):1110-20. doi: 10.1056/NEJMoa065464. PMID 17360989
- [Background] Hideshima T, Podar K, Chauhan D, Ishitsuka K, Mitsiades C, Tai YT, Hamasaki M, Raje N, Hideshima H, Schreiner G, Nguyen AN, Navas T, Munshi NC, Richardson PG, Higgins LS, Anderson KC. p38 MAPK inhibition enhances PS-341 (bortezomib)-induced cytotoxicity against multiple myeloma cells. Oncogene. 2004 Nov 18;23(54):8766-76. doi: 10.1038/sj.onc.1208118. PMID 15480425
- [Background] Shringarpure R, Catley L, Bhole D, Burger R, Podar K, Tai YT, Kessler B, Galardy P, Ploegh H, Tassone P, Hideshima T, Mitsiades C, Munshi NC, Chauhan D, Anderson KC. Gene expression analysis of B-lymphoma cells resistant and sensitive to bortezomib. Br J Haematol. 2006 Jul;134(2):145-56. doi: 10.1111/j.1365-2141.2006.06132.x. PMID 16846475
- [Background] Godfrey J, Benson DM Jr. The role of natural killer cells in immunity against multiple myeloma. Leuk Lymphoma. 2012 Sep;53(9):1666-76. doi: 10.3109/10428194.2012.676175. Epub 2012 Apr 19. PMID 22423650
- [Background] Lawrence T, Natoli G. Transcriptional regulation of macrophage polarization: enabling diversity with identity. Nat Rev Immunol. 2011 Oct 25;11(11):750-61. doi: 10.1038/nri3088. PMID 22025054
- [Background] Ratta M, Fagnoni F, Curti A, Vescovini R, Sansoni P, Oliviero B, Fogli M, Ferri E, Della Cuna GR, Tura S, Baccarani M, Lemoli RM. Dendritic cells are functionally defective in multiple myeloma: the role of interleukin-6. Blood. 2002 Jul 1;100(1):230-7. doi: 10.1182/blood.v100.1.230. PMID 12070032
- [Background] Favaloro J, Brown R, Aklilu E, Yang S, Suen H, Hart D, Fromm P, Gibson J, Khoo L, Ho PJ, Joshua D. Myeloma skews regulatory T and pro-inflammatory T helper 17 cell balance in favor of a suppressive state. Leuk Lymphoma. 2014 May;55(5):1090-8. doi: 10.3109/10428194.2013.825905. Epub 2013 Aug 28. PMID 23865833
- [Background] Rosenberg SA, Restifo NP. Adoptive cell transfer as personalized immunotherapy for human cancer. Science. 2015 Apr 3;348(6230):62-8. doi: 10.1126/science.aaa4967. PMID 25838374
- [Background] Garfall AL, Maus MV, Hwang WT, Lacey SF, Mahnke YD, Melenhorst JJ, Zheng Z, Vogl DT, Cohen AD, Weiss BM, Dengel K, Kerr ND, Bagg A, Levine BL, June CH, Stadtmauer EA. Chimeric Antigen Receptor T Cells against CD19 for Multiple Myeloma. N Engl J Med. 2015 Sep 10;373(11):1040-7. doi: 10.1056/NEJMoa1504542. PMID 26352815
- [Background] Casucci M, Nicolis di Robilant B, Falcone L, Camisa B, Norelli M, Genovese P, Gentner B, Gullotta F, Ponzoni M, Bernardi M, Marcatti M, Saudemont A, Bordignon C, Savoldo B, Ciceri F, Naldini L, Dotti G, Bonini C, Bondanza A. CD44v6-targeted T cells mediate potent antitumor effects against acute myeloid leukemia and multiple myeloma. Blood. 2013 Nov 14;122(20):3461-72. doi: 10.1182/blood-2013-04-493361. Epub 2013 Sep 9. PMID 24016461
- [Background] Shaffer DR, Savoldo B, Yi Z, Chow KK, Kakarla S, Spencer DM, Dotti G, Wu MF, Liu H, Kenney S, Gottschalk S. T cells redirected against CD70 for the immunotherapy of CD70-positive malignancies. Blood. 2011 Apr 21;117(16):4304-14. doi: 10.1182/blood-2010-04-278218. Epub 2011 Feb 8. PMID 21304103
- [Background] Drent E, Groen RW, Noort WA, Themeli M, Lammerts van Bueren JJ, Parren PW, Kuball J, Sebestyen Z, Yuan H, de Bruijn J, van de Donk NW, Martens AC, Lokhorst HM, Mutis T. Pre-clinical evaluation of CD38 chimeric antigen receptor engineered T cells for the treatment of multiple myeloma. Haematologica. 2016 May;101(5):616-25. doi: 10.3324/haematol.2015.137620. Epub 2016 Feb 8. PMID 26858358
- [Background] Drent E, Themeli M, Poels R, de Jong-Korlaar R, Yuan H, de Bruijn J, Martens ACM, Zweegman S, van de Donk NWCJ, Groen RWJ, Lokhorst HM, Mutis T. A Rational Strategy for Reducing On-Target Off-Tumor Effects of CD38-Chimeric Antigen Receptors by Affinity Optimization. Mol Ther. 2017 Aug 2;25(8):1946-1958. doi: 10.1016/j.ymthe.2017.04.024. Epub 2017 May 13. PMID 28506593
- [Background] O'Connell FP, Pinkus JL, Pinkus GS. CD138 (syndecan-1), a plasma cell marker immunohistochemical profile in hematopoietic and nonhematopoietic neoplasms. Am J Clin Pathol. 2004 Feb;121(2):254-63. doi: 10.1309/617D-WB5G-NFWX-HW4L. PMID 14983940
- [Background] Matsui W, Wang Q, Barber JP, Brennan S, Smith BD, Borrello I, McNiece I, Lin L, Ambinder RF, Peacock C, Watkins DN, Huff CA, Jones RJ. Clonogenic multiple myeloma progenitors, stem cell properties, and drug resistance. Cancer Res. 2008 Jan 1;68(1):190-7. doi: 10.1158/0008-5472.CAN-07-3096. PMID 18172311
- [Background] Ramos CA, Savoldo B, Torrano V, Ballard B, Zhang H, Dakhova O, Liu E, Carrum G, Kamble RT, Gee AP, Mei Z, Wu MF, Liu H, Grilley B, Rooney CM, Brenner MK, Heslop HE, Dotti G. Clinical responses with T lymphocytes targeting malignancy-associated kappa light chains. J Clin Invest. 2016 Jul 1;126(7):2588-96. doi: 10.1172/JCI86000. Epub 2016 Jun 6. PMID 27270177
- [Background] Hsi ED, Steinle R, Balasa B, Szmania S, Draksharapu A, Shum BP, Huseni M, Powers D, Nanisetti A, Zhang Y, Rice AG, van Abbema A, Wong M, Liu G, Zhan F, Dillon M, Chen S, Rhodes S, Fuh F, Tsurushita N, Kumar S, Vexler V, Shaughnessy JD Jr, Barlogie B, van Rhee F, Hussein M, Afar DE, Williams MB. CS1, a potential new therapeutic antibody target for the treatment of multiple myeloma. Clin Cancer Res. 2008 May 1;14(9):2775-84. doi: 10.1158/1078-0432.CCR-07-4246. PMID 18451245
- [Background] Chu J, He S, Deng Y, Zhang J, Peng Y, Hughes T, Yi L, Kwon CH, Wang QE, Devine SM, He X, Bai XF, Hofmeister CC, Yu J. Genetic modification of T cells redirected toward CS1 enhances eradication of myeloma cells. Clin Cancer Res. 2014 Aug 1;20(15):3989-4000. doi: 10.1158/1078-0432.CCR-13-2510. Epub 2014 Mar 27. PMID 24677374
- [Background] Ali SA, Shi V, Maric I, Wang M, Stroncek DF, Rose JJ, Brudno JN, Stetler-Stevenson M, Feldman SA, Hansen BG, Fellowes VS, Hakim FT, Gress RE, Kochenderfer JN. T cells expressing an anti-B-cell maturation antigen chimeric antigen receptor cause remissions of multiple myeloma. Blood. 2016 Sep 29;128(13):1688-700. doi: 10.1182/blood-2016-04-711903. Epub 2016 Jul 13. PMID 27412889
- [Background] Rotolo A, Caputo V, Karadimitris A. The prospects and promise of chimeric antigen receptor immunotherapy in multiple myeloma. Br J Haematol. 2016 May;173(3):350-64. doi: 10.1111/bjh.13976. Epub 2016 Mar 8. PMID 26953076
- [Background] Carpenter RO, Evbuomwan MO, Pittaluga S, Rose JJ, Raffeld M, Yang S, Gress RE, Hakim FT, Kochenderfer JN. B-cell maturation antigen is a promising target for adoptive T-cell therapy of multiple myeloma. Clin Cancer Res. 2013 Apr 15;19(8):2048-60. doi: 10.1158/1078-0432.CCR-12-2422. Epub 2013 Jan 23. PMID 23344265
- [Background] Novak AJ, Darce JR, Arendt BK, Harder B, Henderson K, Kindsvogel W, Gross JA, Greipp PR, Jelinek DF. Expression of BCMA, TACI, and BAFF-R in multiple myeloma: a mechanism for growth and survival. Blood. 2004 Jan 15;103(2):689-94. doi: 10.1182/blood-2003-06-2043. Epub 2003 Sep 25. PMID 14512299
- [Background] Ryan MC, Hering M, Peckham D, McDonagh CF, Brown L, Kim KM, Meyer DL, Zabinski RF, Grewal IS, Carter PJ. Antibody targeting of B-cell maturation antigen on malignant plasma cells. Mol Cancer Ther. 2007 Nov;6(11):3009-18. doi: 10.1158/1535-7163.MCT-07-0464. PMID 18025285
- [Background] Xu S, Lam KP. B-cell maturation protein, which binds the tumor necrosis factor family members BAFF and APRIL, is dispensable for humoral immune responses. Mol Cell Biol. 2001 Jun;21(12):4067-74. doi: 10.1128/MCB.21.12.4067-4074.2001. PMID 11359913
- [Background] Matsui W, Huff CA, Wang Q, Malehorn MT, Barber J, Tanhehco Y, Smith BD, Civin CI, Jones RJ. Characterization of clonogenic multiple myeloma cells. Blood. 2004 Mar 15;103(6):2332-6. doi: 10.1182/blood-2003-09-3064. Epub 2003 Nov 20. PMID 14630803
- [Background] Zah E, Lin MY, Silva-Benedict A, Jensen MC, Chen YY. T Cells Expressing CD19/CD20 Bispecific Chimeric Antigen Receptors Prevent Antigen Escape by Malignant B Cells. Cancer Immunol Res. 2016 Jun;4(6):498-508. doi: 10.1158/2326-6066.CIR-15-0231. Epub 2016 Apr 8. PMID 27059623
- [Background] Grada Z, Hegde M, Byrd T, Shaffer DR, Ghazi A, Brawley VS, Corder A, Schonfeld K, Koch J, Dotti G, Heslop HE, Gottschalk S, Wels WS, Baker ML, Ahmed N. TanCAR: A Novel Bispecific Chimeric Antigen Receptor for Cancer Immunotherapy. Mol Ther Nucleic Acids. 2013 Jul 9;2(7):e105. doi: 10.1038/mtna.2013.32. PMID 23839099